CLINICAL TRIAL: NCT04569084
Title: A Phase 3b, Multicenter, Randomized, Double-Blind Study to Evaluate Efficacy and Safety of Oral Edaravone Administered for a Period of 48 Weeks in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Efficacy and Safety Study of Oral Edaravone Administered in Subjects With ALS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility was met.
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-1186-A02; jRCT2031200301 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2019-004256-11 (EudraCT Number)
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: ALS
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT-1186 (Experimental)
  Interventions: Drug: MT-1186
- MT-1186 and Placebo (Experimental)
  Interventions: Drug: MT-1186; Drug: Placebo

INTERVENTIONS:
Drug: MT-1186 — Oral edaravone
  Other Names: Oral edaravone
Drug: Placebo — Oral
  Arms: MT-1186 and Placebo

SUMMARY:
To evaluate and compare the efficacy of two dosing regimens of oral edaravone in subjects with amyotrophic lateral sclerosis (ALS) based on the change in ALS Functional Rating Scale- Revised (ALSFRS-R) score from baseline up to Week 48:

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide a signed and dated informed consent form (ICF) to participate in the study. Subjects must be able (in the judgment of the Investigator) to understand the nature of the study and all risks involved with participation in the study. Subjects must be willing to cooperate and comply with all protocol restrictions and requirements.
2. Subjects will be male or female, ≥ 18 to 75 years of age at the time the ICF is signed.
3. Subjects will be diagnosed with Definite ALS or Probable ALS according to the El Escorial revised criteria for the diagnosis of ALS.
4. Subjects with a baseline score ≥ 2 points on each individual item of the ALSFRS- R at screening and baseline visits.
5. Subjects have a screening and baseline %forced vital capacity (FVC) ≥ 70%.
6. Subjects with 1- to 4-point decline for 8 weeks (±7 days) in ALSFRS-R total score between screening and baseline visits.
7. Subjects whose first symptom of ALS has occurred within 2 years of providing written informed consent.

Exclusion Criteria:

Exclusions Related to Primary Diagnosis

1. Subjects with a history of spinal surgery after the onset of ALS, such as surgery for cervical spondylosis or a herniated disc, or plans for such surgery during the study period.

   Exclusions Related to Other Neurological Disorders (including, but not limited to the following)
2. Subjects with the possibility that the current symptoms may be symptoms of a disease requiring differential diagnosis, such as cervical spondylosis and multifocal motor neuropathy, cannot be ruled out.

   Exclusions Related to General Health or Concomitant Conditions
3. Subjects undergoing treatment for a malignancy.
4. Subjects with a complication that could have a significant effect on efficacy evaluations, such as Parkinson's disease or syndrome, schizophrenia, bipolar disorder, and dementia.
5. Subjects who have the presence or history of any clinically significant (CS) disease (except ALS) that could interfere with the objectives of the study (the assessment of safety and efficacy) or the safety of the subject, as judged by the Investigator.
6. Subjects who are female, of childbearing potential, and pregnant (a positive pregnancy test) or lactating at the screening visit (Visit 1).
7. Subjects of childbearing potential unwilling to use acceptable method of contraception from the screening visit until 3 months after the last dose of study medication. Subjects who are sexually active who do not agree to use contraception during the study period.
8. Subjects who have a significant risk of suicidality. Subjects with any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without a specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the Columbia-Suicide Severity Rating Scale (C-SSRS) within the 3 months before the screening visit.
9. Subjects who have alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevations greater than 2 times the upper limit of normal (ULN) at screening.
10. Subjects with a Glomerular Filtration Rate (GFR) < 30 mL/Min Per 1.73 m2 at screening, using the Larsson Equation.

    Exclusions Related to Medications
11. Subjects with history of hypersensitivity to edaravone, any of the additives or inactive ingredients of edaravone, or sulfites.
12. Subjects with hereditary problems of fructose intolerance (eg, fructose, sucrose, invert sugar, and sorbitol).
13. Subjects who participated in another study and were administered an investigational product within 1 month or 5 half-lives of the investigational agent, whichever is longer, before providing informed consent for the present study.
14. Subjects who have received any previous treatment with edaravone.
15. Subjects who have received stem cell therapy.
16. Subjects who are unable to take their medications orally at baseline (Visit 2).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (95):
- United States (34):
  - St. Joseph's Hospital and Medical Center (SJHMC), Phoenix, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - Woodland Research Northwest, Rogers, Arkansas
  - UCSD Medical Center, La Jolla, California
  - Loma Linda University Health Care - Department of Neurology, Loma Linda, California
  - University California Los Angeles Medical Center (UCLA), Los Angeles, California
  - University of California Irvine (UCI) Health - Women's Healthcare Center, Orange, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - UF Health Cancer Center, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of South Florida (USF) - Carol and Frank Morsani Center for Advanced Health Care (CAHC), Tampa, Florida
  - Emory University - School of Medicine, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Ochsner Center for Primary Care and Wellness, Jefferson, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Lahey Hospital, Burlington, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Neurology Associates, P.C. - Lincoln, Lincoln, Nebraska
  - Las Vegas Clinic, Las Vegas, Nevada
  - Dent Neurologic Institute, Amherst, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Jefferson Weinberg ALS Center, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania
  - University Of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Wesley Neurology Clinic, P.C., Cordova, Tennessee
  - Austin Neuromuscular Center, Austin, Texas
  - Nerve And Muscle Center Of Texas, Houston, Texas
  - The University of Vermont (UVM) and UVM Medical Center National ALS Center of Excellence, Burlington, Vermont
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - St. Luke's Rehabilitation Institute, Spokane, Washington
  - West Virginia University School of Medicine (WVUSoM) - Movement Disorder Clinic, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (10):
  - University of Alberta - Walter C Mackenzie Health Sciences Centre (WCM), Edmonton, Alberta
  - Regional Health Authority B, Fredericton, New Brunswick
  - Health Science Center Mcmaster University, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Odette Cancer Center-Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Recherche Sepmus, Inc, Greenfield Park, Quebec
  - Centre Hospitalier De L'Universite De Montreal (Chum) Notre-Dame Hospital, Montreal, Quebec
  - Montreal Neurological Institute And Hospital, Montreal, Quebec
  - CHU de Quebec-Hopital-Enfant-Jesus, Québec, Quebec
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
- Germany (11):
  - Universitaetsklinikum Wuerzburg, Wuezburg, Germany
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - UKRUB - Berufsgenossenschaftliches Universitatsklinikum Bergmannsheil GmbH - Medizinische Klinik III, Bochum, North Rhine-Westphalia
  - Charite Campus Virchow, Berlin
  - Universitätsklinik Bonn-Motoneuronambulanz, Klinik und Poliklinik für Neurodegenerative Erkrankungen und Gerontopsychiatrie, Bonn
  - Georg-August-Universitaet Goettingen - Universitaetsmedizin Goettingen (UMG), Göttingen
  - Universitaetsklinikum Jena, Jena
  - Klinikum Rechts der Isar der Technischen Universitaet Muenchen, München
  - University Medical Center Rostock, Rostock
  - Universitaets- und Rehabilitationskliniken Ulm, Ulm
  - Deutsche Klinik fuer Diagnostik, Wiesbaden
- Italy (7):
  - Universita degli Studi di Torino - Centro Regionale Esperto Per La Sclerosi Laterale Amiotrofica (CRESLA), Turin, Piedmont
  - Fondazione Serena Onlus - Azienda Ospedaliera Niguarda Ca Granda - Centro Clinico Nemo (Neuro Muscular Omnicentre), Milan
  - Ospedale San Raffaele (HSR) (Istituto Scientifico Universitario San Raffaele), Milan
  - Istituto Nazionale Neurologico Carlo Besta, Milan
  - Istituto Auxologico Italiano - Istituto Di Ricovero e Cura a Carattere Scientifico - Istituto Scientifico Ospedale San Luca, Modena
  - Centro SLA di Palermo, Palermo
  - Policlinico A. Gemelli, Roma
- Japan (26):
  - National Hospital Organization Higashinagoya National Hospital, Meito-ku, Nagoya-shi, Aichi-ken
  - Nagoya University Hospital, Showa-ku, Nagoya, Aichi-ken
  - National Hospital Organization Chibahigashi National Hospital, Chuo-ku, Chiba-shi, Chiba
  - Murakami Karindoh Hospital, Nishi-ku, Fukuoka-shi, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hiroshima University Hospital, Minami-ku, Hiroshima-shi, Hiroshima
  - National Hospital Organization Hokkaido Medical Center, Sapporo, Hokkaido
  - National Hospital Organization Iou National Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Miki-cho, Kita-gun, Kagawa-ken
  - Yokohama City University Hospital, Kanazawa-ku, Yokohama-shi, Kanagawa
  - Kitasato University Hospital, Minami-ku, Sagamihara-city, Kanagawa
  - National Hospital Organization Kumamoto Saishun Medical Center, Koshi-shi, Kumamoto
  - National Hospital Organization Utano National Hospital, Ukyo-ku, Kyoto City, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital, Asahimachidori, Chuo-ku, Niigata-shi, Niigata
  - Kansai Electric Power Hospital, Fukushima-ku, Osaka-shi, Osaka
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka-shi, Osaka
  - Saitama Neuropsychiatric Institute, Chuo-ku, Saitama-shi, Saitama
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - National Hospital Organization Shizuoka Institute of Epilepsy and Neurological Disorders, Aoi-ku, Shizuoka-shi, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Neurological Hospital, Fuchū, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Chiba University Hospital, Chiba
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Switzerland (4):
  - University hospital Bern (Inselspital), Bern, Canton of Bern
  - Hopitaux Universitaires de Geneve (HUG) (Hopital Cantonal), Geneva
  - Neurocenter of Southern Switzerland, Lugano
  - Zentrumsleiter Muskelzentrum/ALS Clinic Kantonsspital St.Gallen Muskelzentrum/ALS Clinic, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rothstein J, Genge A, De Silva S, Zinman L, Chum M, Chio A, Sobue G, Aoki M, Yoshino H, Doyu M, Selness D, Todorovic V, Sasson N, Hirai M, Takahashi F, Salah A, Wamil A, Apple S. Efficacy and Safety of Once Daily Dosing vs. Approved On/Off Dosing of Edaravone Oral Suspension Up to 48 Weeks in Patients With Amyotrophic Lateral Sclerosis (Study MT-1186-A02). Muscle Nerve. 2025 Sep;72(3):433-442. doi: 10.1002/mus.28448. Epub 2025 Jun 6. PMID 40474686

RESULTS

PARTICIPANT FLOW:
Groups:
- Edaravone 105 mg (Once Daily): Oral edaravone 105 mg administered once daily (regimen denoted as Once Daily) in Cycles 1 through 12
- Edaravone 105mg (2 Weeks On/Off ): Oral edaravone 105 mg administered for 14 days, followed by placebo for 14 days in Cycle 1.
  Subsequently, repeat oral edaravone 105 mg administered for 10 days followed by placebo for 18 days (regimen denoted as On/Off) in Cycles 2 through 12
Period: Overall Study
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105mg (2 Weeks On/Off )
Started | 192 | 192
Completed | 125 | 121
Not Completed | 67 | 71
Not completed — Adverse Event | 10 | 14
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 3 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 20 | 21
Not completed — Study terminated by sponsor | 26 | 23
Not completed — Other | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105mg (2 Weeks On/Off ) | Total
Number analyzed (Participants) | 192 | 192 | 384
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 134 | 122 | 256
  65-84 years | 58 | 70 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 139
  Male | 123 | 122 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 183 | 187 | 370
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: CAFS Score at Week 48
Description: CAFS ranks patients' clinical outcomes based on survival time and change in the ALSFRS-R score. To calculate a patient's CAFS, each patient is compared individually to all other patients in the study. The summary score for each patient is the sum of the comparisons ( 1, 0, 1) against all other patients.
  After that, patients' summary scores are ranked. The CAFS rank is 1-383 and a higher CAFS rank indicates a better outcome than does a lower CAFS.
  Since CAFS were calculated using the imputed ALSFRS-R scores with multiple imputation method, and the maximum varies for each simulation, 383 is the maximum possible value of full range for measure of dispersion.
Time Frame: up to 48 Weeks
Population: One subject randomized to the On/Off treatment group was excluded from this analysis because the subject did not receive any study treatment.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105mg (2 Weeks On/Off )
Number analyzed (Participants) | 192 | 191
Units on a scale | 187.2 [4 to 383] | 184.2 [1 to 383]
Statistical Analysis 1: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105mg (2 Weeks On/Off ); Test type: Superiority; p = 0.777, ANCOVA

2. Secondary Outcome: Change From Baseline in % Slow Vital Capacity (SVC) at Week 48
Description: SVC measurements will be conducted in clinic at around the same time of day where possible with the subject in sitting upright position. Subjects should make at least 3 attempts to generate acceptable and reproducible SVC data. The highest value was selected and recorded.
Time Frame: up to 48 Weeks
Population: Those patients reached to Week 48 and conducted SVC assessment.
Measure: Least Squares Mean (Standard Error); unit: percentage of SVC
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105mg (2 Weeks On/Off )
Number analyzed (Participants) | 116 | 117
percentage of SVC | -26.94 (2.45) | -22.15 (2.48)
Statistical Analysis 1: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105mg (2 Weeks On/Off ); Test type: Superiority; p = 0.169, Mixed Model for Repeated Measures (MMRM)

3. Secondary Outcome: Change From Baseline in Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ)40 at Week 48
Description: The ALSAQ-40 is a questionnaire that consists of 40 questions/items with 5 discrete scales: physical mobility, activities of daily living and independence, eating and drinking, communication, emotional reactions, ranging from 0 (best health as assessed by the scale) to 100 (worse health as assessed by the measure).
Time Frame: up to 48 Weeks
Population: Those patients reached to Week 48 and conducted ALSAQ-40 assessment.
Measure: Least Squares Mean (Standard Error); unit: Point
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105mg (2 Weeks On/Off )
Number analyzed (Participants) | 128 | 125
Point | 2.35 (0.25) | 1.79 (0.25)

4. Secondary Outcome: Time to Death, Tracheostomy or Permanent Assisted Mechanical Ventilation (≥ 23 Hours/Day)
Time Frame: up to 48 Weeks
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105mg (2 Weeks On/Off )
Number analyzed (Participants) | 192 | 192
Months | NA [NA to NA] — The median survival time to death, tracheostomy, or PAMV at 50% survival probability timepoint could not be calculated (K-M analysis) in either group due to the low number of events (Once Daily group: 11 events; On/Off group: 17 events), resulting in 181 and 175 censored observations in respective group. | NA [NA to NA] — The median survival time to death, tracheostomy, or PAMV at 50% survival probability timepoint could not be calculated (K-M analysis) in either group due to the low number of events (Once Daily group: 11 events; On/Off group: 17 events), resulting in 181 and 175 censored observations in respective group.

5. Secondary Outcome: Time to Death or PAMV (≥ 23 Hours/Day)
Time Frame: up to 48 Weeks
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105mg (2 Weeks On/Off )
Number analyzed (Participants) | 192 | 192
Months | NA [NA to NA] — The median survival time to death or PAMV at 50% survival probability timepoint could not be calculated (K-M analysis) in either group due to the low number of events (Once Daily group: 10 events; On/Off group: 17 events). | NA [NA to NA] — The median survival time to death or PAMV at 50% survival probability timepoint could not be calculated (K-M analysis) in either group due to the low number of events (Once Daily group: 10 events; On/Off group: 17 events).

6. Secondary Outcome: Time to Death
Time Frame: up to 48 Weeks
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105mg (2 Weeks On/Off )
Number analyzed (Participants) | 192 | 192
Months | NA [NA to NA] — The median survival time to death at 50% survival probability timepoint could not be calculated (K-M analysis) in either group due to the low number of events (Once Daily group: 9 events; On/Off group: 16 events). | NA [NA to NA] — The median survival time to death at 50% survival probability timepoint could not be calculated (K-M analysis) in either group due to the low number of events (Once Daily group: 9 events; On/Off group: 16 events).

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: The safety analysis set (SAF) is defined as all randomized subjects who received at least 1 dose of study medication. One subject randomized to the on/off treatment group was excluded from the arm because the subject did not receive any study treatment. Therefore, serious, and other AE were analyzed by SAF which is 2weeks on/off Group: 191, whereas the number at Risk for All-Cause Mortality is Randomized set which is 2weeks on/off Group: 192, considering the definition of ClinicalTrials.gov.
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105mg (2 Weeks On/Off )
All-Cause Mortality (participants affected / at risk) | 9/192 | 16/192
Serious Adverse Events (participants affected / at risk) | 52/192 | 55/191
Other Adverse Events (participants affected / at risk) | 118/192 | 131/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edaravone 105 mg (Once Daily) (N=192) | Edaravone 105mg (2 Weeks On/Off ) (N=191)
Cardiac arrest (Cardiac disorders) | 1 | 2
Benign familial pemphigus (Congenital, familial and genetic disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 16 | 15
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 1
Sudden death (General disorders) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 4 | 4
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Coronavirus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 1
Swallow study (Investigations) | 0 | 1
Vital capacity decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 5
Syncope (Nervous system disorders) | 1 | 2
Embedded device (Product Issues) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Gastrostomy (Surgical and medical procedures) | 3 | 0
Jejunostomy (Surgical and medical procedures) | 0 | 1
Artery dissection (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edaravone 105 mg (Once Daily) (N=192) | Edaravone 105mg (2 Weeks On/Off ) (N=191)
Constipation (Gastrointestinal disorders) | 24 | 27
Diarrhoea (Gastrointestinal disorders) | 20 | 14
Dysphagia (Gastrointestinal disorders) | 11 | 12
Fatigue (General disorders) | 12 | 10
Oedema peripheral (General disorders) | 10 | 9
COVID-19 (Infections and infestations) | 24 | 26
Nasopharyngitis (Infections and infestations) | 11 | 8
Contusion (Injury, poisoning and procedural complications) | 17 | 14
Fall (Injury, poisoning and procedural complications) | 36 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 10
Headache (Nervous system disorders) | 15 | 9
Depression (Psychiatric disorders) | 9 | 10
Insomnia (Psychiatric disorders) | 11 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 8
Rash (Skin and subcutaneous tissue disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT04569084/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT04569084/SAP_001.pdf